CLINICAL TRIAL: NCT04635033
Title: Safety and Tolerance of an Intermittent Intervention in MS Patients
Brief Title: Intermittent Hypoxia Intervention in MS Patients
Acronym: MSHYPE
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Christoph Heesen, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: MS HYPE Pilot
Record Dates: First submitted 2020-10-22; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: 2 hours of reduced FiO2 (11-15%) in the inspired air, 2-3x/week, 3 months

SUMMARY:
This observational cohort study investigates the safety and feasibility of an intermittent hypoxia intervention in multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* confirmed MS (all types of MS)
* ability to come to the outpatient clinic 2-3x/week for 3 months
* EDSS ≤ 6.5
* inconspicuous medical examination
* inconspicuous ECG

Exclusion Criteria:

* relapse in the last 3 months
* EDSS progression in the last 6 months
* pregnancy
* contraindication for MRI
* severe heart disease
* severe asthma, COPD
* cancer
* severe cognitive deficits
* chronic headache
* renal insufficiency
* anaemia (Hb < 10 g/dl)
* insulin-dependent diabetes mellitus
* severe vascular stenosis
* former episodes of severe high mountain sickness
* cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MS patients with all types of MS
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Lake Louise Score (LLS) | Change of mean LLS before vs. after 1 hour vs. after 2 hours of each session
  Tolerance by measuring the development of acute mountain sickness during the sessions Score 3 to 5 = mild AMS Score 6 or more = severe AMS

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  MS impairment measurement with a score ranging from 0.0 (normal neurological exam) to 10.0 (death due to MS)
Timed 25-Foot Walk (T25-FW) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Quantitative mobility and leg function performance test based on a timed 25-walk
6 minute walking test (6MWT) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Maximum distance in 6 minutes
9-Hole-Peg-Test (9 HPT) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Quantitative test of upper extremity function
Verbal learning and memory test (VLMT) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Rapid and delayed recall
Symbol Digit Modalities Test (SDMT) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Test for concentration and decision making
Brief Visuospatial Memory Test-Revised (BVMT-R) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Test for visuospatial memory
Frenchay Activities Index (FAI) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Measure of instrumental activities of daily living (IADL)
Fatigue Scale Motor Cognition (FSMC) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Measure MS-related cognitive and motor fatigue in MS
  * 43 Mild Fatigue
  * 53 Medium Fatigue
  * 63 Severe Fatigue
Beck Depression Inventory (BDI) | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Measure severity of depression
MRI Lesions | Baseline, at the end of the intervention (after 3 months)
  T2 and Gd enhancing T1 lesions
Brain atrophy | Baseline, at the end of the intervention (after 3 months)
  MRI
Immune cell subsets | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  FACS analysis
Heart rate | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  bpm by pulsoxymeter
Blood pressure | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  mmHg
Heart rate | During every session (2hours/session)
  bpm by pulsoxymeter
Oxygen saturation | During every session (2hours/session)
  measured by pulsoxymeter
Blood sugar | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  mg/dl in the blood sample
Blood count | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Hb, Hct, Leucocytes, Lymphocytes, Thrombocytes, Neutrophils in th blood sample
Erythropoetin | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  blood sample
Liver enzymes | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  GOT, GPT, GGT (blood sample)
Kidney enzyme | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Creatinine (blood sample)
NFL | Baseline, 4 weeks after starting the intervention, at the end of the intervention (after 3 months)
  Neurofilament light chain (serum)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, INIMS, Hamburg, Germany